CLINICAL TRIAL: NCT01876459
Title: Rate of Alpha-synuclein in Cerebrospinal Fluid to Differentiate Patient With Alzheimer's Disease From Those With Lewy Body Disease.
Brief Title: Alpha-synuclein in Cerebrospinal Fluid to Differentiate Alzheimer's Disease From Lewy Body Disease.
Acronym: AlphaLewyMa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 5330; N° IDRCB 2012-A00992-41 (Other: ANSM)
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: "Alzheimer's Disease" and "Lewy Body Disease"
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Disease | interventions — Spinal Puncture; Neuropsychological Tests

ARMS (2):
- "Alzheimer's Disease" arm (Other): Patient with Alzheimer's disease
  Interventions: Other: MRI; Procedure: lumbar puncture; Behavioral: neuropsychological tests
- "Lewy Body Disease" arm (Other): Patient with Lewy Body Disease
  Interventions: Other: MRI; Procedure: lumbar puncture; Behavioral: neuropsychological tests

INTERVENTIONS:
Other: MRI
Procedure: lumbar puncture
Behavioral: neuropsychological tests

SUMMARY:
Patients with memory disorders are experiencing different trends which are difficult to predict. Moreover, the distinction between Lewy body disease and Alzheimer's disease is not easy as both diseases can present similar symptoms. Nowadays, routine examinations exist and can improve the diagnosis but there are not specific enough of one of those two pathologies.

Lewy body disease is characterized by the presence of particular structures in patient's brain, called "Lewy body", composed of a protein called "alpha-synuclein". The aim of this study is to measure the rate of alpha-synuclein in cerebrospinal fluid. This measurement could allow us to differentiate patient with Alzheimer's disease from those with Lewy body disease.

ELIGIBILITY:
Inclusion Criteria:

* At least 45 years of age
* Subject agrees to participate in the study
* Subject meets the criteria Dubois et al., 2007. for diagnosis of probable AD.
* Subject with a syndromic presentation of mild cognitive impairment or mild dementia
* Subject has a study partner who is able to provide accurate information about the patient
* Subject affiliated to a social security scheme

Exclusion Criteria:

* Patient who meets both AD and Lewy Body disease criteria
* Contraindications to lumbar puncture
* Contraindications to an MRI scan
* Subject who is not affiliated to a social security scheme
* Subject under guardianship or curatorship
* Subject under judicial protection
* Subject refuses to participate in the study
* Subject has evidence of clinically relevant neurological disorder (fronto-temporal dementia, brain tumor, stroke, …) that led to persistent cognitive disorders
* Subject has evidence of clinically relevant psychiatric disorders (schizophrenia, major depression, …)
* Pregnant or attempting to become pregnant women
* Subject's vision and audition is sufficient for neuropsychological tests's assessment, based on the investigator's judgment.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
rate of alpha-synuclein in cerebrospinal fluid | Day one.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, Hôpital de Hautepierre, France

REFERENCES:
- [Derived] Gabriel V, Chabran E, Sourty M, Cretin B, Philippi N, Muller C, Anthony P, Demuynck C, Loureiro de Sousa P, Botzung A, Sanna L, Bousiges O, Blanc F. Salience and frontoparietal network impairments across disease stages in dementia with Lewy bodies: A comparative functional MRI study with Alzheimer's disease. J Alzheimers Dis. 2025 Dec;108(3):1398-1409. doi: 10.1177/13872877251386844. Epub 2025 Oct 17. PMID 41105629
- [Derived] Querry M, Botzung A, Sourty M, Chabran E, Sanna L, Loureiro de Sousa P, Cretin B, Demuynck C, Muller C, Ravier A, Schorr B, Philippi N, Blanc F. Functional Connectivity Changes Associated With Depression in Dementia With Lewy Bodies. Int J Geriatr Psychiatry. 2025 Mar;40(3):e70058. doi: 10.1002/gps.70058. PMID 40011213
- [Derived] Sainsily-Cesarus A, Schmitt E, Landre L, Botzung A, Rauch L, Demuynck C, Philippi N, de Sousa PL, Mutter C, Cretin B, Martin-Hunyadi C, Blanc F. Dementia with Lewy bodies and gait neural basis: a cross-sectional study. Alzheimers Res Ther. 2024 Jul 30;16(1):170. doi: 10.1186/s13195-024-01539-z. PMID 39080741
- [Derived] Bousiges O, Cretin B, Muller C, Botzung A, Sanna L, Anthony P, Philippi N, Demuynck C, Blanc F. Involvement of ApoE4 in dementia with Lewy bodies in the prodromal and demented stages: evaluation of the Strasbourg cohort. Geroscience. 2024 Apr;46(2):1527-1542. doi: 10.1007/s11357-023-00883-6. Epub 2023 Aug 31. PMID 37653269
- [Derived] Mendes A, Noblet V, Mondino M, Loureiro de Sousa P, Manji S, Archenault A, Casanovas M, Bousiges O, Philippi N, Baloglu S, Rauch L, Cretin B, Demuynck C, Martin-Hunyadi C, Blanc F. Association of cerebral microbleeds with cerebrospinal fluid Alzheimer-biomarkers and clinical symptoms in early dementia with Lewy bodies. Int J Geriatr Psychiatry. 2021 Jun;36(6):851-857. doi: 10.1002/gps.5485. Epub 2020 Dec 26. PMID 33300151
- [Derived] Bousiges O, Philippi N, Lavaux T, Perret-Liaudet A, Lachmann I, Schaeffer-Agalede C, Anthony P, Botzung A, Rauch L, Jung B, de Sousa PL, Demuynck C, Martin-Hunyadi C, Cretin B, Blanc F. Differential diagnostic value of total alpha-synuclein assay in the cerebrospinal fluid between Alzheimer's disease and dementia with Lewy bodies from the prodromal stage. Alzheimers Res Ther. 2020 Sep 29;12(1):120. doi: 10.1186/s13195-020-00684-5. PMID 32993772